CLINICAL TRIAL: NCT06262386
Title: Utilizing Perioperative Variation Trends of Circulating Tumor Cells and Tumor Pathological Characteristics as a Combined Relapse Prediction Model for Resectable Non-Small Cell Patients - a Prospective Clinical Feasibility Trial
Brief Title: Combined Relapse Prediction Model for Resectable Non-Small Cell Patients - a Prospective Clinical Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202202172B0
Record Dates: First submitted 2023-09-22; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer; Relapse/Recurrence
Keywords: Circulating tumor cell; resectable non-small cell lung cancer; Early relapse
MeSH Terms: conditions — Lung Neoplasms; Recurrence; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient at risk for disease relapse after surgery (Experimental): 1. we utilized a relapse prediction model that combined perioperative variation trends of circulating tumor cells and pathologic characteristics that were collated with relapse
     1. circulating tumor cell variation trend: difference between the CTC count on post-operation day 3 and day 1; difference between the CTC count on post-operation day 3 and post-operation
     2. pathologic staging 0-1a/ 1b-4
  2. patient with high relapse for relapse
     * Adjuvant was recommended as NCCN guidelines recommended
  Interventions: Drug: Cisplatin based chemottherapy

INTERVENTIONS:
Drug: Cisplatin based chemottherapy — adjuvant therapy for high risk patient

SUMMARY:
For patients with lung cancer who have undergone tumor resection, early relapse significantly impacts survival. However, there are currently no reliable screening or imaging tools available to identify patients at risk of early relapse. To address this clinical challenge, many studies have focused on understanding the clinicopathologic characteristics associated with an increased risk of early relapse. Despite these efforts, we can identify patients at risk but cannot pinpoint which individuals will actually experience early relapse. Studies on adjuvant therapy have shown improved survival in cases of more advanced disease but have not demonstrated a reduction in early relapse rates.

In our preliminary analysis of previous study data, we observed that patients with a smaller reduction in circulating tumor cells (CTCs) within the first three days after surgery, followed by an increase on the third-day post-operation, are more likely to experience early relapse during regular monitoring. This pattern may be indicative of minimal residual disease. By combining trends in circulating tumor cell variations with pathologic characteristics, we aim to select patients for adjuvant therapy who are at high risk of developing early relapse.

The objective of our study is to employ screening based on circulating tumor cell dynamics and pathologic features to identify patients likely to experience early relapse and to assess the effectiveness of adjuvant therapy in these cases.

DETAILED DESCRIPTION:
For patients with resectable lung cancer, anatomic resection alongside mediastinal lymph node dissection is pivotal in removing all tumor tissue visible on imaging from the patient's body. Despite these efforts, early relapse remains a significant issue. Literature review shows that the early relapse rate varies between 8 to 10%, potentially due to undetectable occult metastasis by imaging modalities, suggesting the presence of minimal residual disease or tumor cells evading the primary site. Limitations in imaging, such as the slice thickness in computed tomography (CT) scans, which range from 0.375 to 0.5 centimeters, can render tumors smaller than the slice thickness invisible. Similarly, tumors smaller than 0.5 cm may not accumulate sufficient F18-Deoxyglucose to be detectable in positron emission tomography (PET) scans. Additionally, tumor cells may migrate to extrapulmonary sites via lymphatic drainage or circulation.

Survival studies have predominantly focused on the pathologic TNM stage, which aggregates different disease presentations with similar survival outcomes. However, the heterogeneity inherent in pathology may help in identifying patients prone to relapse. From a tumor biology perspective, tumor cells may detach from surrounding tissues, becoming more invasive and entering the bloodstream. Circulating tumor cells (CTCs) have been recognized early in cancer stages and are correlated with treatment response, tumor genetic alterations, and survival. Research has combined CT tumor size and CTCs in a malignancy prediction model for suspicious pulmonary lesions, highlighting that CTCs can rebound in patients experiencing early relapse, indicating occult metastases or minimal residual disease.

Systemic adjuvant therapy is considered the best approach to minimize disease relapse in resectable lung cancer patients. Although many studies have sought to identify patients at risk of relapse to improve survival, the presence of intrapulmonary (N1) or mediastinal (N2) lymph node invasion significantly affects survival in non-small cell lung cancer patients. Even tumors smaller than 1 cm carry a risk of lymph node metastases, with respective risks for cT1a, cT1b, and cT1c tumors reported as 3.8%, 16.3%, and 19.6%. Therefore, patients with tumors larger than 1 cm are recommended adjuvant therapy due to the high risk of lymph node involvement. Adjuvant chemotherapy is advised for patients with stages 1b to 3a, showing a 5.4% survival benefit by the fifth postoperative year, although this benefit diminishes in subsequent years. This could be due to adjuvant therapy being administered based on the pathologic stage rather than the likelihood of relapse. Tumor heterogeneity might also influence the response to different therapeutic regimens. Molecular profiling of tumors has identified mutations predicting responses to targeted therapies and elucidated drug resistance mechanisms, offering more precise treatments and improving survival. Targeted and immune therapies have shown improved survival in specific tumor subgroups.

This study aims to utilize trends in CTC variations as a screening tool to identify patients at risk of relapse and prescribe adjuvant therapy to evaluate the therapeutic efficacy and survival impact of CTCs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who presented with resectable disease ( Clinical stage 1a to 3a)
2. Patients who received tumor resection

Exclusion Criteria:

1. Pathologic stage greater than stage 3b or 4
2. Pathologic stage less than stage 1a1
3. Could not complete treatment course
4. Could not receive blood sampling for CTC (circulating tumor cell) or regular surveillance

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of proposed relapse prediction model | follow up in 3 month-interval
  1. Utilized the enrolled patients to testify proposed relapse prediction model
  2. Calculated Positive prediction rate, Negative prediction rate, accuracy
  3. Goal: high positive prediction rate, lower negative prediction rate, high accuracy
early relapse rate | follow up in 3 month-interval
  1. adjuvant therapy based on proposed relapse prediction model
     * calculate the early relapse rate (relapse within 3 years)
  2. utilized historical cohort as historical control (cohort that utilized to establish proposed relapse prediction model
     * adjuvant therapy based on TNM stage
     * calculate the early relapse rate (relapse within 3 years)
     * follow up Chest CT/ CTC in 3-month interval

SECONDARY OUTCOMES:
Overall surveival | follow up in 3 month-interval
  Goal: difference of overall survival among patients with relapse risk
  1. treatment based on proposed relapse prediction model
  2. calculate the overall survival
  3. utilized historical cohort as historical control ( cohort that utilized to establish proposed relapse prediction model
     * treatment based on TNM stage
     * calculate the overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yang Wu, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Ching-Yang Wu, Taoyuan, Taiwan

REFERENCES:
- [Result] Wu CY, Fu JY, Wu CF, Liu YH, Hsieh MJ, Wu YC, Yang CT, Tsai YH. Pathologic Stage of Nonsmall Cell Lung Cancer Patients Presenting as Resectable Cases After Neoadjuvant Therapy Did Not Predict the Prognosis. Medicine (Baltimore). 2015 Oct;94(40):1. doi: 10.1097/MD.0000000000001700. PMID 26448022
- [Result] Boedeker KL, Cooper VN, McNitt-Gray MF. Application of the noise power spectrum in modern diagnostic MDCT: part I. Measurement of noise power spectra and noise equivalent quanta. Phys Med Biol. 2007 Jul 21;52(14):4027-46. doi: 10.1088/0031-9155/52/14/002. Epub 2007 Jun 8. PMID 17664593
- [Result] Sun F, Xi J, Zhan C, Yang X, Wang L, Shi Y, Jiang W, Wang Q. Ground glass opacities: Imaging, pathology, and gene mutations. J Thorac Cardiovasc Surg. 2018 Aug;156(2):808-813. doi: 10.1016/j.jtcvs.2018.02.110. Epub 2018 Apr 13. PMID 29753514
- [Result] Funama Y, Awai K, Liu D, Oda S, Yanaga Y, Nakaura T, Kawanaka K, Shimamura M, Yamashita Y. Detection of nodules showing ground-glass opacity in the lungs at low-dose multidetector computed tomography: phantom and clinical study. J Comput Assist Tomogr. 2009 Jan-Feb;33(1):49-53. doi: 10.1097/RCT.0b013e31815e6291. PMID 19188784
- [Result] Dahlbom M, Hoffman EJ, Hoh CK, Schiepers C, Rosenqvist G, Hawkins RA, Phelps ME. Whole-body positron emission tomography: Part I. Methods and performance characteristics. J Nucl Med. 1992 Jun;33(6):1191-9. PMID 1597738
- [Result] Nolop KB, Rhodes CG, Brudin LH, Beaney RP, Krausz T, Jones T, Hughes JM. Glucose utilization in vivo by human pulmonary neoplasms. Cancer. 1987 Dec 1;60(11):2682-9. doi: 10.1002/1097-0142(19871201)60:113.0.co;2-h. PMID 3499969
- [Result] Brown RS, Leung JY, Kison PV, Zasadny KR, Flint A, Wahl RL. Glucose transporters and FDG uptake in untreated primary human non-small cell lung cancer. J Nucl Med. 1999 Apr;40(4):556-65. PMID 10210213
- [Result] Pieterman RM, van Putten JW, Meuzelaar JJ, Mooyaart EL, Vaalburg W, Koeter GH, Fidler V, Pruim J, Groen HJ. Preoperative staging of non-small-cell lung cancer with positron-emission tomography. N Engl J Med. 2000 Jul 27;343(4):254-61. doi: 10.1056/NEJM200007273430404. PMID 10911007
- [Result] Gupta GP, Massague J. Cancer metastasis: building a framework. Cell. 2006 Nov 17;127(4):679-95. doi: 10.1016/j.cell.2006.11.001. PMID 17110329
- [Result] Fidler IJ. The pathogenesis of cancer metastasis: the 'seed and soil' hypothesis revisited. Nat Rev Cancer. 2003 Jun;3(6):453-8. doi: 10.1038/nrc1098. PMID 12778135
- [Result] Carbone DP, Salmon JS, Billheimer D, Chen H, Sandler A, Roder H, Roder J, Tsypin M, Herbst RS, Tsao AS, Tran HT, Dang TP. VeriStrat classifier for survival and time to progression in non-small cell lung cancer (NSCLC) patients treated with erlotinib and bevacizumab. Lung Cancer. 2010 Sep;69(3):337-40. doi: 10.1016/j.lungcan.2009.11.019. Epub 2009 Dec 29. PMID 20036440
- [Result] Maheswaran S, Sequist LV, Nagrath S, Ulkus L, Brannigan B, Collura CV, Inserra E, Diederichs S, Iafrate AJ, Bell DW, Digumarthy S, Muzikansky A, Irimia D, Settleman J, Tompkins RG, Lynch TJ, Toner M, Haber DA. Detection of mutations in EGFR in circulating lung-cancer cells. N Engl J Med. 2008 Jul 24;359(4):366-77. doi: 10.1056/NEJMoa0800668. Epub 2008 Jul 2. PMID 18596266
- [Result] O'Flaherty JD, Gray S, Richard D, Fennell D, O'Leary JJ, Blackhall FH, O'Byrne KJ. Circulating tumour cells, their role in metastasis and their clinical utility in lung cancer. Lung Cancer. 2012 Apr;76(1):19-25. doi: 10.1016/j.lungcan.2011.10.018. Epub 2011 Dec 29. PMID 22209049
- [Result] Nieva J, Wendel M, Luttgen MS, Marrinucci D, Bazhenova L, Kolatkar A, Santala R, Whittenberger B, Burke J, Torrey M, Bethel K, Kuhn P. High-definition imaging of circulating tumor cells and associated cellular events in non-small cell lung cancer patients: a longitudinal analysis. Phys Biol. 2012 Feb;9(1):016004. doi: 10.1088/1478-3975/9/1/016004. Epub 2012 Feb 3. PMID 22306961
- [Result] Wu CY, Lee CL, Wu CF, Fu JY, Yang CT, Wen CT, Liu YH, Liu HP, Hsieh JC. Circulating Tumor Cells as a Tool of Minimal Residual Disease Can Predict Lung Cancer Recurrence: A longitudinal, Prospective Trial. Diagnostics (Basel). 2020 Mar 6;10(3):144. doi: 10.3390/diagnostics10030144. PMID 32155787
- [Result] Wu CF, Wu CY, Fu JY, Wang CW, Liu YH, Hsieh MJ, Wu YC. Prognostic value of metastatic N1 lymph node ratio and angiolymphatic invasion in patients with pathologic stage IIA non-small cell lung cancer. Medicine (Baltimore). 2014 Oct;93(20):e102. doi: 10.1097/MD.0000000000000102. PMID 25365403
- [Result] Fu JY, Wan YL, Huang TY, Wu CF, Liu YH, Hsieh MJ, Wu YC, Wu CY. Correction: Correlation between image characteristics and pathologic findings in non small cell lung cancer patients after anatomic resection. PLoS One. 2019 Feb 12;14(2):e0212461. doi: 10.1371/journal.pone.0212461. eCollection 2019. PMID 30753242
- [Result] Sonobe M, Date H, Wada H, Okubo K, Hamakawa H, Teramukai S, Matsumura A, Nakagawa T, Sumitomo S, Miyamoto Y, Okumura N, Takeo S, Kawakami K, Aoki M, Kosaka S; The Japan-Multinational Trial Organization. Prognostic factors after complete resection of pN2 non-small cell lung cancer. J Thorac Cardiovasc Surg. 2013 Oct;146(4):788-95. doi: 10.1016/j.jtcvs.2013.04.043. Epub 2013 Jun 27. PMID 23810113
- [Result] Misthos P, Sepsas E, Athanassiadi K, Kakaris S, Skottis I. Skip metastases: analysis of their clinical significance and prognosis in the IIIA stage of non-small cell lung cancer. Eur J Cardiothorac Surg. 2004 Apr;25(4):502-8. doi: 10.1016/j.ejcts.2004.01.025. PMID 15037262
- [Result] Schuchert MJ, Normolle DP, Awais O, Pennathur A, Wilson DO, Luketich JD, Landreneau RJ. Factors influencing recurrence following anatomic lung resection for clinical stage I non-small cell lung cancer. Lung Cancer. 2019 Feb;128:145-151. doi: 10.1016/j.lungcan.2018.12.026. Epub 2018 Dec 26. PMID 30642447
- [Result] Lee G, Lee HY, Jeong JY, Han J, Cha MJ, Lee KS, Kim J, Shim YM. Clinical impact of minimal micropapillary pattern in invasive lung adenocarcinoma: prognostic significance and survival outcomes. Am J Surg Pathol. 2015 May;39(5):660-6. doi: 10.1097/PAS.0000000000000399. PMID 25724001
- [Result] Cha MJ, Lee HY, Lee KS, Jeong JY, Han J, Shim YM, Hwang HS. Micropapillary and solid subtypes of invasive lung adenocarcinoma: clinical predictors of histopathology and outcome. J Thorac Cardiovasc Surg. 2014 Mar;147(3):921-928.e2. doi: 10.1016/j.jtcvs.2013.09.045. Epub 2013 Nov 4. PMID 24199757
- [Result] Matsuoka Y, Yurugi Y, Takagi Y, Wakahara M, Kubouchi Y, Sakabe T, Haruki T, Araki K, Taniguchi Y, Nakamura H, Umekita Y. Prognostic Significance of Solid and Micropapillary Components in Invasive Lung Adenocarcinomas Measuring </=3 cm. Anticancer Res. 2016 Sep;36(9):4923-30. doi: 10.21873/anticanres.11058. PMID 27630350
- [Result] Kato H, Ichinose Y, Ohta M, Hata E, Tsubota N, Tada H, Watanabe Y, Wada H, Tsuboi M, Hamajima N, Ohta M; Japan Lung Cancer Research Group on Postsurgical Adjuvant Chemotherapy. A randomized trial of adjuvant chemotherapy with uracil-tegafur for adenocarcinoma of the lung. N Engl J Med. 2004 Apr 22;350(17):1713-21. doi: 10.1056/NEJMoa032792. PMID 15102997
- [Result] Douillard JY, Rosell R, De Lena M, Carpagnano F, Ramlau R, Gonzales-Larriba JL, Grodzki T, Pereira JR, Le Groumellec A, Lorusso V, Clary C, Torres AJ, Dahabreh J, Souquet PJ, Astudillo J, Fournel P, Artal-Cortes A, Jassem J, Koubkova L, His P, Riggi M, Hurteloup P. Adjuvant vinorelbine plus cisplatin versus observation in patients with completely resected stage IB-IIIA non-small-cell lung cancer (Adjuvant Navelbine International Trialist Association [ANITA]): a randomised controlled trial. Lancet Oncol. 2006 Sep;7(9):719-27. doi: 10.1016/S1470-2045(06)70804-X. PMID 16945766
- [Result] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Result] Arriagada R, Dunant A, Pignon JP, Bergman B, Chabowski M, Grunenwald D, Kozlowski M, Le Pechoux C, Pirker R, Pinel MI, Tarayre M, Le Chevalier T. Long-term results of the international adjuvant lung cancer trial evaluating adjuvant Cisplatin-based chemotherapy in resected lung cancer. J Clin Oncol. 2010 Jan 1;28(1):35-42. doi: 10.1200/JCO.2009.23.2272. Epub 2009 Nov 23. PMID 19933916
- [Result] Wood SL, Pernemalm M, Crosbie PA, Whetton AD. Molecular histology of lung cancer: from targets to treatments. Cancer Treat Rev. 2015 Apr;41(4):361-75. doi: 10.1016/j.ctrv.2015.02.008. Epub 2015 Feb 20. PMID 25825324
- [Result] Felip E, Altorki N, Zhou C, Csoszi T, Vynnychenko I, Goloborodko O, Luft A, Akopov A, Martinez-Marti A, Kenmotsu H, Chen YM, Chella A, Sugawara S, Voong D, Wu F, Yi J, Deng Y, McCleland M, Bennett E, Gitlitz B, Wakelee H; IMpower010 Investigators. Adjuvant atezolizumab after adjuvant chemotherapy in resected stage IB-IIIA non-small-cell lung cancer (IMpower010): a randomised, multicentre, open-label, phase 3 trial. Lancet. 2021 Oct 9;398(10308):1344-1357. doi: 10.1016/S0140-6736(21)02098-5. Epub 2021 Sep 20. PMID 34555333
- [Result] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177
- [Result] Duan GC, Zhang XP, Wang HE, Wang ZK, Zhang H, Yu L, Xue WF, Xin ZF, Hu ZH, Zhao QT. Circulating Tumor Cells as a Screening and Diagnostic Marker for Early-Stage Non-Small Cell Lung Cancer. Onco Targets Ther. 2020 Mar 4;13:1931-1939. doi: 10.2147/OTT.S241956. eCollection 2020. PMID 32184628
- [Result] Schwartz LH, Litiere S, de Vries E, Ford R, Gwyther S, Mandrekar S, Shankar L, Bogaerts J, Chen A, Dancey J, Hayes W, Hodi FS, Hoekstra OS, Huang EP, Lin N, Liu Y, Therasse P, Wolchok JD, Seymour L. RECIST 1.1-Update and clarification: From the RECIST committee. Eur J Cancer. 2016 Jul;62:132-7. doi: 10.1016/j.ejca.2016.03.081. Epub 2016 May 14. PMID 27189322
- [Result] Thornblade LW, Mulligan MS, Odem-Davis K, Hwang B, Waworuntu RL, Wolff EM, Kessler L, Wood DE, Farjah F. Challenges in Predicting Recurrence After Resection of Node-Negative Non-Small Cell Lung Cancer. Ann Thorac Surg. 2018 Nov;106(5):1460-1467. doi: 10.1016/j.athoracsur.2018.06.022. Epub 2018 Jul 19. PMID 30031845
- [Result] Okumura Y, Tanaka F, Yoneda K, Hashimoto M, Takuwa T, Kondo N, Hasegawa S. Circulating tumor cells in pulmonary venous blood of primary lung cancer patients. Ann Thorac Surg. 2009 Jun;87(6):1669-75. doi: 10.1016/j.athoracsur.2009.03.073. PMID 19463575
- [Result] Su PJ, Wu MH, Wang HM, Lee CL, Huang WK, Wu CE, Chang HK, Chao YK, Tseng CK, Chiu TK, Lin NM, Ye SR, Lee JY, Hsieh CH. Circulating Tumour Cells as an Independent Prognostic Factor in Patients with Advanced Oesophageal Squamous Cell Carcinoma Undergoing Chemoradiotherapy. Sci Rep. 2016 Aug 17;6:31423. doi: 10.1038/srep31423. PMID 27530152